CLINICAL TRIAL: NCT01527747
Title: Effects of Dipeptidyl Peptidase-4 Inhibition With Saxagliptin on Fasting and Postprandial Triglyceride Concentrations
Brief Title: Effects of DPP-4 Inhibition on Triglycerides
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, P. Barton Duell, M.D., Director, Lipid-Atherosclerosis Laboratory, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CV181-142
Record Dates: First submitted 2012-01-31; First posted 2012-02-07 (Estimated); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes; Hypertriglyceridemia
Keywords: Type 2 Diabetes; Hypertriglyceridemia; dipeptidyl peptidase-4 (DPP-4); glucagon-like peptide-1 (glp-1)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertriglyceridemia | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo arm
  Interventions: Drug: Saxagliptin
- Saxagliptin (Experimental): Active drug arm
  Interventions: Drug: Saxagliptin

INTERVENTIONS:
Drug: Saxagliptin — 5 mg daily
  Other Names: Onglyza

SUMMARY:
The purpose of this study is to test the effects of saxagliptin, a treatment for diabetes, on fasting and post-meal blood triglyceride (blood fat) levels.

DETAILED DESCRIPTION:
This study is designed to help us understand the effects of DPP-4 inhibition on triglyceride levels before and after eating.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide signed written informed consent
* Men and women aged 18-80 years
* Type 2 diabetes (as defined by the ADA - see reference 18)
* Baseline HgbA1c between 6.5% and 8%; HgbA1c 7.5-8.0% among subjects taking sulfonylureas
* Baseline plasma triglyceride concentration between 200 and 700 mg/dl
* Stable diabetes medication regimen for at least 12 weeks prior to study entry
* Taking a statin for at least 8 weeks, unless statin therapy is contraindicated or intolerable
* Treatment with other lipid-lowering medications only if the dose has been stable for > 8 weeks.
* Non-smoker
* Body mass index < 45.0 kg/m2
* BP < 140/85
* Normal serum TSH and free T4 concentrations (hypothyroid subjects taking a stable replacement dose of levothyroxine will be allowed if they are biochemically euthyroid)
* Subjects will otherwise be healthy
* Women of child-bearing potential must be willing to use reliable contraception, as defined by our IRB, throughout the study (There are currently no FDA recommended restrictions on the use of saxagliptin in sexually active men, or requirements for contraception in their wives or sexual partners)
* Able and willing to complete study procedures

Exclusion Criteria:

* Transaminase concentrations > 2 times the ULN. (Mild elevations of AST and ALT will be allowed up to 2x ULN at baseline if there is no evidence of viral hepatitis or intrinsic liver disease. Since many of these subjects may have some degree of hepatic steatosis, a key intervention is the implementation of treatment to lower glucose and triglycerides)
* Estimated creatinine clearance < 60 ml/min
* Microalbumin-creatinine ratio > 120
* Alcohol consumption > 1 drink daily in women and > 2 drinks daily in men
* Pancreatitis within the preceding 6 months
* Type 1 diabetes
* History of diabetic ketoacidosis (DKA)
* Cardiovascular disease (CAD, stroke, PVD)
* Known human immunodeficiency virus (HIV) infection
* Viral hepatitis
* Pregnancy or lactation
* A current diagnosis of active non-dermatologic cancer
* Other life-threatening illness
* History of small bowel resection or gastric bypass surgery
* Use of glucocorticoid medications, beta blockers, thiazide diuretics, excess alcohol intake (beta-blockers and thiazide diuretic will be allowed, if necessary, if the dose has been stable for > 12 weeks prior to study entry and the dose will remain stable throughout the study. Complete exclusion of these drugs would exclude a substantial proportion of diabetic patients)
* Use of systemic cytochrome P450 3A4 (CYP 3A4/5) inhibitors such as ketaconazole, atazanavir, clarithromycin, indinavir, itraconazole, nefazodone, nelfinavir, ritonavir, saquinavir and telithromycin.
* Current enrollment in another research study or use of any investigational drug within 90 days of study entry
* Other medical conditions that may interfere with participation in the study, in the opinion of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-01; Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in fasting and postprandial triglyceride concentrations | baseline, 6 weeks
  Comparison of 6 weeks of placebo vs 6 weeks of saxagliptin

SECONDARY OUTCOMES:
Changes in glycemia | baseline, 6 weeks
  Comparison of 6 weeks of placebo vs 6 weeks of saxagliptin

CONTACTS AND LOCATIONS:
Overall Officials: P Barton Duell, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No